CLINICAL TRIAL: NCT01398046
Title: Effects of Gastric pH on the Pharmacokinetics of Dasatinib in Healthy Volunteers
Brief Title: Effects of Gastric pH on the Pharmacokinetics of Dasatinib
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: Dasatinib-63-03
Record Dates: First submitted 2011-07-05; First posted 2011-07-20 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Healthy
Keywords: dasatinib; betaine; betaine hydrochloride; pharmacokinetics; healthy volunteer
MeSH Terms: interventions — Dasatinib; Rabeprazole; Betaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dasatinib (Active Comparator)
  Interventions: Drug: Dasatinib
- Dasatinib plus Rabeprazole (Experimental)
  Interventions: Drug: Dasatinib plus Rabeprazole
- Dasatinib plus Rabeprazole AND Betaine Hydrochloride (Experimental)
  Interventions: Drug: Dasatinib plus Rabeprazole AND Betaine Hydrochloride

INTERVENTIONS:
Drug: Dasatinib — dasatinib (100mg) PO x1
  Arms: Dasatinib
Drug: Dasatinib plus Rabeprazole — Rabeprazole (20mg) PO twice daily (Days 1-3); Dasatinib (100mg) PO x1 (Day 4)
  Arms: Dasatinib plus Rabeprazole
Drug: Dasatinib plus Rabeprazole AND Betaine Hydrochloride — Rabeprazole (20mg) PO twice daily (Days 1-3); Betaine Hydrochloride (1500mg) PO x1 AND Dasatinib (100mg) PO x1 on Day 4
  Arms: Dasatinib plus Rabeprazole AND Betaine Hydrochloride

SUMMARY:
The goal of this study is to evaluate the ability of a natural supplement (betaine hydrochloride) to affect the absorption of dasatinib in healthy volunteers. The investigators predict that betaine hydrochloride will increase the absorption of dasatinib, in volunteers pre-treated with proton-pump inhibitors (PPIs).

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18-59 years of age
* Healthy adult with no active medical problems or significant chronic diseases as determined by the study doctor based on history, physical exam and laboratory evaluations
* BMI between 18.5-30 kg/m2
* Taking no medications 2 weeks before and during the study enrollment, including drugs of abuse, prescription or over-the-counter (OTC) medications (except acetaminophen)
* Subjects able to maintain adequate birth control during the study independent of hormonal contraceptive use
* Be able to provide written informed consent and comply with requirements of the study
* Avoid eating grapefruit and drinking grapefruit juice from 7 days before the first study day until the completion of the entire study
* Abstinence from alcoholic beverages, caffeinated beverages and orange juice from 3pm the night before a study day until completion of that study day
* Fast from food and beverages at least 8 hours prior to medication dosing
* Be able to read, speak, and understand English

Exclusion Criteria:

* Subjects with a history of gastrointestinal disease including gastroesophageal reflux disease, gastritis, peptic ulcer disease, or dyspepsia
* Subjects with a fasting gastric pH of > 4 (i.e. hypochlorhydria)
* Subjects with a history of dysphagia, achalasia, or difficulty swallowing capsules, tablets, or pills
* Subjects on prescription or chronic over-the-counter (OTC) medications (including hormonal contraceptives)
* Subjects with known allergies to rabeprazole or any other proton pump inhibitors (PPI's) or betaine hydrochloride
* Subjects who smoke tobacco
* Subjects with ongoing alcohol or illegal drug use
* Subjects who are pregnant, lactating, or attempting to conceive
* Subjects unable to maintain adequate birth control during the study

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2011-08; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Area-Under-the Concentration Curve from zero-to-twenty two hours (AUC,0-22) of Dasatinib | Day 4
  The primary outcome measure will be dasatinib area-under-the-concentration curve (AUC) values from zero-to-twenty two (0-22) hours. Values from Experiemntal Arms of the study (Dasatinib plus Rabeprazole; Dasatinib plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (dasatinib alone) and tested for statistical significance.
Area-Under-the Concentration Curve from zero-to-infinity (AUC,0-inf) of Dasatinib | Day 4
  The primary outcome measure will be dasatinib area-under-the-concentration curve (AUC) values from zero-to-infinite time (0-inf). Values from Experiemntal Arms of the study (Dasatinib plus Rabeprazole; Dasatinib plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (dasatinib alone) and tested for statistical significance.

SECONDARY OUTCOMES:
Maximum Concentration of Dasatinib | Day 4
  The maximum plasma concentration (Cmax) will also be measured. Values from Experiemntal Arms of the study (Dasatinib plus Rabeprazole; Dasatinib plus Rabeprazole AND Betaine Hydrochloride) will be compared against the active comparator (Dasatinib alone) and tested for statistical significance.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Z Benet, Ph.D, Principal Investigator — University of California, San Francisco; Lynda Frassetto, M.D., Principal Investigator — University of California, San Francisco
Locations (1):
- Clinical Research Center, UCSF, San Francisco, California, United States

REFERENCES:
- [Derived] Yago MR, Frymoyer AR, Smelick GS, Frassetto LA, Budha NR, Dresser MJ, Ware JA, Benet LZ. Gastric reacidification with betaine HCl in healthy volunteers with rabeprazole-induced hypochlorhydria. Mol Pharm. 2013 Nov 4;10(11):4032-7. doi: 10.1021/mp4003738. Epub 2013 Sep 10. PMID 23980906